CLINICAL TRIAL: NCT06323473
Title: Maitake for Integrative Cancer Care: An Open Label, Uncontrolled Trial in People on Systemic Cancer Therapy
Brief Title: Maitake for Integrative Cancer Care
Acronym: Maitake
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Maitake001
Record Dates: First submitted 2024-02-27; First posted 2024-03-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: Chemotherapy; Maitake; Integrative Care; Integrative Medicine; Targeted Therapy; Neutrophil
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Uncontrolled single arm clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Maitake given alongside systemic chemotherapy and/or CD4/6 inhibitors
  Interventions: Dietary Supplement: Black Maitake Prothera

INTERVENTIONS:
Dietary Supplement: Black Maitake Prothera — Mushroom extract; liquid
  Other Names: Grifola Fondosa; Maitake

SUMMARY:
Maitake is an edible mushroom that is used for both its nutritional and medicinal properties. Human and animal studies have shown Maitake may help improve immune function; however, its effectiveness in people with cancer is not clear. The investigators aim to measure if Maitake has any immunomodulatory effects when given alongside conventional systemic cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years of age)
2. Confirmed cancer diagnosis through biopsy or radiologic imaging
3. Undergoing systemic treatment with either chemotherapy or CD4/6 inhibitors
4. Currently receiving cancer treatment in Ontario, Canada

Exclusion Criteria:

1. Hematologic cancers
2. Previously received any mushroom supplement within 6 months prior to enrolment
3. Allergy to mushrooms or mushroom products
4. Diagnosis of diabetes
5. Currently taking hypoglycemic or anticoagulant medications
6. Currently receiving immune checkpoint inhibitors
7. Unable to attend in in-person visits in either Ottawa or Toronto
8. Any reason which, under the discretion of the Qualified Investigator or delegate, would preclude the patient from participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Changes in absolute neutrophil count | Baseline, week 4, week 8, week 12, week 16
  The investigators will assess within-person changes in blood neutrophils throughout the study. Normal limit is 2.00 - 7.50 x 10^9/L, where a higher neutrophil count will be considered an improvement. Values above the normal limit will be excluded due to the potential of infection.

SECONDARY OUTCOMES:
Incidence of febrile neutropenia | Baseline, week 4, week 8, week 12, week 16
  Febrile neutropenia is defined as absolute neutrophil count < 1.0 x 10^9/L and temperature > 38.3 degrees Celsius.
Change in neutrophil to lymphocyte ratio (NLR) | Baseline, week 4, week 8, week 12, week 16
  Higher NLRs have been associated with poorer cancer prognosis. The investigators will assess within-person changes in NLR where a lower value in considered favourable. Values of neutrophils or lymphocytes outside the normal limit will be excluded due to the potential for infection.
Change in platelet to lymphocyte ratio (PLR) | Baseline, week 4, week 8, week 12, week 16
  Higher PLRs have been associated with poorer cancer prognosis. The investigators will assess within-person changes in PLR where a lower value in considered favourable. Values of lymphocytes outside the normal limit will be excluded due to the potential for infection.
Change in high-sensitivity C-reactive protein (CRP) | Baseline, week 4, week 8, week 12, week 16
  CRP is a measure of inflammation. Higher levels of inflammation have been linked with poorer cancer prognosis. The investigators will assess within-person changes in CRP as a measure of systemic inflammation. Values less than 10 mg/mL are considered normal, with lower values being favourable.
Changes in Quality of Life | Baseline, week 4, week 8, week 12, week 16
  QOL will be evaluated using the European Organization for Research and Treatment of Cancer's Quality of Life Questionnaire C30 (EORTC QLQ C30), version 3.0, a validated tool for analyzing health-related QOL in patients with cancer participating in clinical trials. The questionnaire incorporates five functional scales, (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a global health status, and a number of single items assessing additional symptoms. Scores range from 0-100 for each item. For functional scales and global health status, a higher score is favourable. For all symptom scales, a lower score is favourable.
Changes in hemoglobin A1c (HbA1c) | Baseline, week 4, week 8, week 12, week 16
  HbA1c is a measure of blood glucose management, an item which is thought to be modulated by Maitake. The investigators will evaluate within-person changes in this metric as a measure of safety. Values below 5.7% are considered normal, with lower values being favourable.
Incidence of adverse events | 16 weeks
  The investigators will collect any adverse events experienced by participants per the common terminology criteria for adverse events (CTCAE) version 5.0.
Incidence of dose reductions or delays in systemic therapy | 16 weeks.
  The investigators will assess the frequency of dose delays or reductions in chemotherapy or CD4/6 inhibitors during the 16-week study period. Dose reductions or delays in treatment can negatively impact outcomes; not having reductions or delays is favourable.
Addition of new medications to combat neutropenia | 16 weeks
  The investigators will assess the incidence of participants requiring new medications (e.g., granulocyte colony-stimulating factor) prescribed to combat neutropenia throughout the 16-week study period. The addition of new medications can cause adverse effects and potentially delay other conventional treatments. The absence of additional medication is considered favourable.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Junek, MD, Principal Investigator — Centre for Health Innovation
Locations (2):
- Canada (2):
  - The Centre for Health Innovation, Ottawa, Ontario
  - Canadian College of Naturopathic Medicine - Integrative Cancer Centre, Toronto, Ontario